CLINICAL TRIAL: NCT02333812
Title: Prevalence of Malignant and Premalignant Lesions in the Head & Neck in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0318-14-HMO-CTIL
Record Dates: First submitted 2014-09-17; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-09

CONDITIONS: COPD, HEAD&NECK CANCER,SCREENING
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- copd patients: Adult patients with COPD
  Interventions: Other: Stroboscopic nasopharyngeal laryngoscopy
- healthy smokers: Adult patients with smoking history and no clinical manifestation of COPD who will be recruited form the institute of pulmonary medicine and the otolaryngology outpatient clinic.
  Interventions: Other: Stroboscopic nasopharyngeal laryngoscopy
- Adult patients with lung disease unrelated to smoking: Adult patients with lung disease unrelated to smoking
  Interventions: Other: Stroboscopic nasopharyngeal laryngoscopy

INTERVENTIONS:
Other: Stroboscopic nasopharyngeal laryngoscopy
  Groups: copd patients
Other: Stroboscopic nasopharyngeal laryngoscopy
  Groups: healthy smokers
Other: Stroboscopic nasopharyngeal laryngoscopy
  Groups: Adult patients with lung disease unrelated to smoking

SUMMARY:
Head and neck cancers usually occur in patients who have a history of long tobacco use. Chronic obstructive pulmonary disease (COPD) is a chronic progressive disease of the airways and lung parenchyma that is also associated with exposure to tobacco. COPD and head & neck cancer share a common environmental risk factor in cigarette smoke exposure. the investigators hypothesize that patients with chronic lung disease related to smoking have a higher risk to develop cancer in the head and neck.

The investigators designed a study to assess the prevalence of cancer and pre-cancer disease in the head & neck in patients with chronic lung disease. the investigators will examine patients with and without a history of smoking and chronic lung disease in order to determine the prevalence of head and neck cancer in the different groups. The patients who will be included in the study will undergo comprehensive evaluation of their lung function and voice performance.

This study is a joint effort of the Pulmonology Institute and the Department of Otolaryngology, Head & Neck Surgery in Israel and the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

1. group of adult COPD patients.
2. Adult patients with smoking history and no clinical manifestation of COPD who will be recruited form the institute of pulmonary medicine and the otolaryngology outpatient clinic.
3. Adult patients with lung disease unrelated to smoking, i.e. bronchial asthma who will be recruited from the institute of pulmonary medicine

Exclusion Criteria:

1. Patients with an acute disease or COPD exacerbation
2. Pregnant patients
3. Patients who were intubated ≤3 months prior to inclusion
4. Patients with a medical history of surgical intervention in the upper airway
5. Patients with a medical history of malignant disease in the upper airway
6. Patients who underwent radiotherapy of head and neck

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group of adult COPD patients will be recruited from the Institute of Pulmonary medicine patient pool and referred for further evaluation in the Voice and Swallowing disorders outpatient Clinic in Hadassah University Medical Center.The study group will be compared to two control group:
  2. Adult patients with smoking history and no clinical manifestation of COPD who will be recruited form the institute of pulmonary medicine and the otolaryngology outpatient clinic.
  3. Adult patients with lung disease unrelated to smoking, i.e. bronchial asthma who will be recruited from the institute of pulmonary medicine
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the primary outcome measure is the number of patients with malignant tumors and pre-malignant lesions of the head & neck | participants will be followed for the duration of hospital stay, an expected average of one week
  prevalence of malignant tumors and pre-malignant lesions of the head & neck in general, and the larynx in particular, is significantly increased in the COPD patient population in comparison to patients with history of smoking without clinical presentation of COPD and patients with no history of smoking.